CLINICAL TRIAL: NCT01301937
Title: Phase III Clinical Trial for Mucosal or Mucocutaneous Leishmaniasis. Comparison Between the Standard and Alternative Antimonial Schemes
Brief Title: Low Antimonial Dosage in American Mucosal Leishmaniasis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, ASchubach, Senior Researcher, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: low dosage ML
Record Dates: First submitted 2011-02-20; First posted 2011-02-23 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Mucosal Leishmaniasis; Mucocutaneous Leishmaniasis
Keywords: Mucosal Leishmaniasis; Leishmania braziliensis; Meglumine Antimoniate; Treatment Effectiveness; Controlled Clinical Trials, Randomized
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous | interventions — Meglumine Antimoniate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High continuous dose (Active Comparator): Meglumine antimoniate 20 mg/kg/day for 30 continuous days
  Interventions: Drug: Meglumine antimoniate
- Low continuous dose (Active Comparator): Meglumine antimoniate 5 mg/kg/day for up to 120 continuous days according to clinical cure
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Meglumine antimoniate — Meglumine antimoniate (Aventis, São Paulo, Brazil) is stored and ministered under actual conditions employed by the health services in Brazil. Each patient will be included in one of two treatment groups with meglumine antimoniate IM:
  1. High continuous dose: 20 mg/kg/day for 30 continuous days.
  2. Low continuous dose 5 mg/kg/day for up to 120 continuous days.
  There will be no cross-over between the groups for the purpose of this study. The data from those patients who require permanent discontinuation of a scheme will be assessed in the group that were randomized, ie, by intention to treat
  Arms: High continuous dose, Low continuous dose
  Other Names: Glucantime

SUMMARY:
"Phase III clinical trial for mucosal or mucocutaneous leishmaniasis. Equivalence between the standard and alternative schemes with meglumine antimoniate" has begun in October 2008 at the Laboratory of Leishmaniasis Surveillance at Evandro Chagas Clinical Research Institute (IPEC), FIOCRUZ, aiming to compare efficacy and safety of the standard recommended schedule with an alternative regimen of meglumine antimoniate (MA) in the treatment of mucosal or mucocutaneous leishmaniasis (ML or MCL)). It is a study with blind evaluation by the doctors and the responsible for statistical analysis. Patients diagnosed with Ml or MCL, eligible for the trial, are randomly allocated into one of the schemes with meglumine antimoniate and monitored before, during and after it. There is no single regimen applicable to all forms of leishmaniasis around the world. Therapeutic regimens applied to treat people living in other geographic areas result in mixed outcomes. Ideally, the most appropriate regimens should be established for each endemic area, based on its efficacy, toxicity, difficulties of administration and cost. Given the problems and limitations of the use of pentavalent antimonials at 20 mg / kg / day, a less toxic alternative regimen with 5mg/kg/day, continuous up to the cure deserves to be better evaluated. Treatment must lead to the healing of mucosal lesions and prevent late scarring tissues and disabilities development. The indication of high doses of MA is based on the evidence that there could be induction of resistance with use of subdoses. However, clinical studies with extended follow-up in Rio de Janeiro have suggested that regular low MA doses (5mg / kg / day) in a systemic way may constitute an effective scheme, achieving cure rates similar to higher dose, with lower toxicity, ease of implementation and lower cost. Published studies on efficacy and safety of alternative schemes with meglumine antimoniate failed to provide conclusive results, for various methodological biases. The need to compare the effectiveness and safety between treatment schemes with meglumine antimoniate currently recommended in Brazil for the treatment of ML or MCL and an alternative scheme with low dose of antimony is the motive for this study in Rio de Janeiro.

DETAILED DESCRIPTION:
1. Introduction. Pentavalent antimonials are first line drugs for the treatment of leishmaniasis. WHO and Brazilian Ministry of Health recommend treating patients with mucosal (ML) or mucocutaneous leishmaniasis (MCL) with doses of 20mg/kg/day, intramuscularly or intravenously, for a period of three to four weeks. In the Reference Centre on Leishmaniasis - IPEC - FIOCRUZ, the dose of 5mg/kg/day IM has been effective and well tolerated in the treatment. ML is treated for 30 continuous or intermittent days, in series of 10 days interspersed with periods of 10 days without medication, up to 12 series of treatment (120 medication days), with a lower incidence of adverse effects and lower treatment dropout rates. The evolution of the lesions is usually similar to that observed with continuous treatment. In all cases patients should be monitored with clinical examination, electrocardiogram, blood count, liver function, renal and pancreatic tests. Some side effects can be observed, although they not necessarily lead to discontinuation of treatment: arthralgia, myalgia, anorexia, abdominal pain, rash, fever, headache, edema, and herpes zoster. Electrocardiographic abnormalities most frequent are heart rhythm and ventricular repolarization disturbances: flattening or inversion of T wave and corrected QT space widening.
2. Background: Ideally, the most appropriate antimoniate therapeutic regimens should be established for each endemic area, based on their efficacy and toxicity, without ignoring the difficulties of administration and cost. The treatment of ML or MCL must achieve the healing of mucosal lesions and prevention of severe scarring of mucosal tissues and consequent disabilities. The recognition, recommendation and acceptance of new regimens should be preceded by demonstration of their superiority to currently recommended treatments. We aim to compare the effectiveness and safety among treatment schemes with meglumine antimoniate currently recommended in Brazil for the treatment of ATL and an alternative scheme with low doses of antimony.
3. Objectives. 3.1. General Objective. To compare the effectiveness and safety of meglumine antimoniate at a dose of 20 mg/kg/day for 30 days or 5 mg continuous up to 120 days, in the treatment of patients with ML or MCL.

   3.2. Specific Objectives. 1. To compare the frequencies of epithelialization and reduction of mucosal infiltration (assessed on days 30, 120, 150 from the beginning of the treatment) between the two groups. 2. To compare the frequencies of good late therapeutic response (maintenance of epithelialization, with total regression of infiltration and no re-emergence of a skin lesion) between the two groups, up to two years. 3. To compare the frequency and severity of adverse clinical, laboratory and electrocardiogram effects between the two groups, controlling for age above or below 60 years. 4. To compare the time in days until the epithelialization and reduction of infiltration of the lesions between the two groups, according to the nasal, oropharyngeal or laryngeal location.
4. Subjects and methods.

4. 1. Study design: Controlled clinical trial with standard and alternative treatment, randomized, double-blind, phase III.

4.2. Description of interventions: Meglumine antimoniate (Aventis, São Paulo, Brazil) is stored and ministered under actual conditions employed by the health services in Brazil. A single lot of medication will be used in all patients. Each patient will be included in one of two treatment groups with meglumine antimoniate IM: 1) 20mg / kg / day for 30 continuous days. Patients with remaining active lesions in the day 120 from the beginning of the treatment will be re-treated with the same regimen. 2) 5mg / kg / day continuous until the epithelization and resolution of mucosal infiltration, respecting the limit of 120 days of treatment.

There will be no cross-over between the groups for the purpose of this study. The data from those patients who require permanent discontinuation of a scheme will be assessed in the group that were randomized, ie, by intention to treat.

4.3. Sampling plan. 4.3.1 Sample size. The comparison of the effectiveness between the two schemes will probably reveal superiority of the alternative scheme (continuous low dose) for the following outcomes: 1) frequency of good initial response (epithelialization and resolution of mucosal infiltration) on day 150. 2) frequency of good late response (maintenance of epithelialization and total regression of infiltration) up to 2 years.

We considered the significance level of 5% and 80% power to calculate the sample sizes needed to compare the groups. Initially, a 76-total of patients will be required (38 patients in each group) to compare the standard group with the alternative group.

4.4 Allocation strategy (randomization). Eligible individuals who agree to participate (by signing an informed consent) will be randomly assigned to one of the two treatment groups, according to order of arrival, until the completion of the groups.

4.5. Eligibility Criteria (see item: Eligibility Criteria). 4.6. Outcomes. 4.6.1 Effectiveness Outcome: Definition: 1. Initial therapeutic response - presence or not of complete epithelization of all lesions until day 150. 2. Late therapeutic response in mucosal leishmaniasis: maintenance of epithelialization and total regression of the infiltration up to 2 years.

4.6.2 Safety Outcomes (adverse events): definition, intensity and relationship to study drug. Adverse events (AE) are considered as any events, adverse or unexpected, evidenced by the investigator or reported by the patients, beginning during the use of the drug or within 30 days after stopping it. The investigation of AE will be made by spontaneous recall and questioned by a physician in a standardized form every 10 days during the medication and in day 30 after completion of treatment. All EA should be monitored until their disappearance.

The classification of the severity of adverse events (clinical, laboratory and electrocardiographic) will take place according to "AIDS Table for Grading Severity of Adult Adverse Experiences, 1992". The causal relationship to study drug (= AE) will be evaluated by the investigator and classified as follows: a) Definite (Highly Likely); b) Probable; c) Possible; d) Remote (Probably not); e) Definitely not.

4.7. Medications allowed. There will be no restrictions on the use of symptomatic medications and for other diseases except those listed in the exclusion criteria.

4.8. Management of adverse effects. The AE will be noted in the appropriate form and shall contain: a description of the adverse effect, its intensity, relation with the investigated drug, start date, completion date, duration and conduct taken.

4.9. Masking. We chose to perform the measurements of outcomes of interest (effectiveness) and adverse events (security) by a physician who is not aware of what is the regimen used by the patient. It is intended to minimize measurement biases of the different outcomes according to treatment regimen to which each patient belongs. The results of laboratory tests are provided by the clinical pathology laboratory without information about the treatment group. The manager of the database will preserve the secrecy of this information by coding the groups for analysis for the epidemiologist (s).

4.10. Criteria for definitive discontinuation of study treatment: a) Interruption driven by clinical, laboratory or electrocardiographic AE Grade 4; b) Interruption exceeding 10 days attributed to clinical, laboratory or electrocardiographic adverse event Grade <3; c) Spontaneous cessation of the use of prescribed medication beyond five consecutive doses, due to fault of the administration (noncompliance).

4.11. Criteria for study withdrawal: a) definitive interruption of treatment; b) pregnancy; c) introduction of immunosuppressive or potentially toxic drugs; d) intercurrent disease, unrelated to study drug, but with manifestations equivalent or superior to clinical grade 3 AE; e) poor initial or late therapeutic response; f) patient abandonment to continue the study.

4.12. Procedures for confidentiality break. The randomization codes used for allocation of numbering and allocation of patients may be revealed in cases of necessity of the study.

4.13. Monitoring the study. The parameters (outcomes) of effectiveness and safety will be monitored according to the timetable for implementation. The principal investigator and coordinators will supervise the field work, controlling for quality deviation and this Protocol. Important items to be monitored: adhesion to the Protocol (follow-up losses will be minimized through active search), appropriate records of outcomes and adverse events; adequacy of stored products; quality of procedures for laboratory tests; minimization of missing data; periodic transmission of data for data entry. Written reports of field will be retained for consideration by the committees. Serious adverse events will be reported to the Ethical Committee and perhaps decision to interrupt the test will be made. External Committee: a committee of outside monitoring of the trial shall be constituted , consisting of three members, experts in the treatment of leishmaniasis and execution of clinical trials. The committee will carry out audits of documentation and activities relevant to the clinical trial, controlling for possible protocol breaks.

4.14 Control of storage of medications. The ampoules required for complete treatment of the whole sample will be stored in IPEC Pharmacy. A trained professional team will include the patients, in day 1 consultation, following the randomization list.

4.15. Data Analysis Plan. Data analysis will be carried out following the principle of intention to treat. The data from those patients who require permanent discontinuation of a scheme will be analyzed according to the group for what they had been allocated initially, not being re-assigned to another group to resumption of treatment (no cross-over between the groups for the purposes of this study). We will describe the simple frequencies of categorical variables and measures of central tendency and dispersion of continuous quantitative variables for each antimony scheme. The proportion of dichotomous outcome of presence or absence of good early and late therapeutic response with the alternative regimen will be compared to the standard one through chi-square test, and the days until the extent of epithelialization and reduction of infiltration of lesions by nasal, oropharyngeal or laryngeal location will be studied through survival time analysis between the two groups (log-rank statistic). If necessary, nonparametric tests will be used. Effectiveness and safety will be also evaluated through relative risk (RR), absolute risk reduction (ARR) and relative risk reduction (RRR).

5. Ethical considerations. 6.1 Risks and benefits. The main potential benefit of this test is the possibility of subsidizing the use of lower doses of antimony, potentially less toxic and less costly. The risks consist of general adverse events, which will be thoroughly scrutinized and treated. This project was submitted to the Ethics in Research Committee (CEP/IPEC) and National Ethics in Research Council (CONEP). All patients sign an informed consent approved by CEP/IPEC. This project follows the recommendations of the National Health Council.

5.2. Informed consent. In plain language and explaining the objectives, risks, benefits and identifying those responsible for research.

6. Expected Results. We hope the different schemes are equivalent in effectiveness, and with diverse toxicities.

7. Financial support. This project is supported in part with funds approved by MCT/CNPq / MS-SCTIE-DECIT 25/2006.

ELIGIBILITY:
Inclusion Criteria:

* Mucosal or mucocutaneous leishmaniasis with parasitological diagnosis by one or more of the following methods: direct examination (imprint), histopathology, culture, immunohistochemistry, or PCR.

Exclusion Criteria:

* Women who do not use contraceptives or do it badly
* Pregnant women
* Children under 13 years
* Previous antimonial treatment for LM
* Immunosuppressive therapy (steroids, cancer chemotherapy) or medicines for tuberculosis or leprosy.
* Presence of altered baseline clinical adverse effect level equivalent to > G3
* Presence of altered basal laboratory adverse effect level equivalent to > G2
* Presence of baseline electrocardiographic changes equivalent to an adverse effect level > G4 and / or baseline QTc > 0.46 ms (equivalent to AE level G1)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2008-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of meglumine antimoniate in the treatment of mucosal leishmaniasis | 6 years
  This study is designed to evaluate the efficacy of high and low doses of meglumine antimoniate in the treatment of mucosal or mucocutaneous leishmaniasis.

SECONDARY OUTCOMES:
Safety of meglumine antimoniate in the treatment of mucosal leishmaniasis | 6 years
  This study is designed to evaluate the safety of hig and low doses of meglumine antimoniate in the treatment of mucosal or mucocutaneous leishmaniasis.

CONTACTS AND LOCATIONS:
Overall Officials: Armando O. Schubach, MD, PhD, Study Director — IPEC/FIOCRUZ
Locations (1):
- Oswaldo Cruz Foundation - IPEC/FIOCRUZ, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antezana G, Zeballos R, Mendoza C, Lyevre P, Valda L, Cardenas F, Noriega I, Ugarte H, Dedet JP. Electrocardiographic alterations during treatment of mucocutaneous leishmaniasis with meglumine antimoniate and allopurinol. Trans R Soc Trop Med Hyg. 1992 Jan-Feb;86(1):31-3. doi: 10.1016/0035-9203(92)90427-e. PMID 1566297
- [Background] de Azeredo-Coutinho RB, Mendonca SC. An intermittent schedule is better than continuous regimen of antimonial therapy for cutaneous leishmaniasis in the municipality of Rio de Janeiro, Brazil. Rev Soc Bras Med Trop. 2002 Sep-Oct;35(5):477-81. doi: 10.1590/s0037-86822002000500009. PMID 12621667
- [Background] Chulay JD, Spencer HC, Mugambi M. Electrocardiographic changes during treatment of leishmaniasis with pentavalent antimony (sodium stibogluconate). Am J Trop Med Hyg. 1985 Jul;34(4):702-9. doi: 10.4269/ajtmh.1985.34.702. PMID 2992303
- [Background] Deps PD, Viana MC, Falqueto A, Dietze R. [Comparative assessment of the efficacy and toxicity of N-methyl-glucamine and BP88 sodium stibogluconate in the treatment of localized cutaneous leishmaniasis]. Rev Soc Bras Med Trop. 2000 Nov-Dec;33(6):535-43. doi: 10.1590/s0037-86822000000600004. Portuguese. PMID 11175583
- [Background] Hepburn NC, Nolan J, Fenn L, Herd RM, Neilson JM, Sutherland GR, Fox KA. Cardiac effects of sodium stibogluconate: myocardial, electrophysiological and biochemical studies. QJM. 1994 Aug;87(8):465-72. PMID 7922300
- [Background] Hepburn NC, Siddique I, Howie AF, Beckett GJ, Hayes PC. Hepatotoxicity of sodium stibogluconate therapy for American cutaneous leishmaniasis. Trans R Soc Trop Med Hyg. 1994 Jul-Aug;88(4):453-5. doi: 10.1016/0035-9203(94)90432-4. PMID 7570843
- [Background] Marzochi MC, Marzochi KB. Tegumentary and visceral leishmaniases in Brazil: emerging anthropozoonosis and possibilities for their control. Cad Saude Publica. 1994;10 Suppl 2:359-75. doi: 10.1590/s0102-311x1994000800014. Epub 2004 Mar 19. PMID 15042226
- [Background] McBride MO, Linney M, Davidson RN, Weber JN. Pancreatic necrosis following treatment of leishmaniasis with sodium stibogluconate. Clin Infect Dis. 1995 Sep;21(3):710. doi: 10.1093/clinids/21.3.710. No abstract available. PMID 8527590
- [Background] Oliveira Neto MP, Schubach A, Araujo ML, Pirmez C. High and low doses of antimony (Sbv) in American cutaneous leishmaniasis. A five years follow-up study of 15 patients. Mem Inst Oswaldo Cruz. 1996 Mar-Apr;91(2):207-9. doi: 10.1590/s0074-02761996000200016. PMID 8736092
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, da Costa SC, Pirmez C. Intralesional therapy of American cutaneous leishmaniasis with pentavalent antimony in Rio de Janeiro, Brazil--an area of Leishmania (V.) braziliensis transmission. Int J Dermatol. 1997 Jun;36(6):463-8. doi: 10.1046/j.1365-4362.1997.00188.x. PMID 9248897
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, Goncalves-Costa SC, Pirmez C. A low-dose antimony treatment in 159 patients with American cutaneous leishmaniasis: extensive follow-up studies (up to 10 years). Am J Trop Med Hyg. 1997 Dec;57(6):651-5. doi: 10.4269/ajtmh.1997.57.651. PMID 9430521
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, Goncalves-Costa SC, Pirmez C. Treatment of American cutaneous leishmaniasis: a comparison between low dosage (5 mg/kg/day) and high dosage (20 mg/kg/day) antimony regimens. Pathol Biol (Paris). 1997 Jun;45(6):496-9. PMID 9309267
- [Background] Ribeiro AL, Drummond JB, Volpini AC, Andrade AC, Passos VM. Electrocardiographic changes during low-dose, short-term therapy of cutaneous leishmaniasis with the pentavalent antimonial meglumine. Braz J Med Biol Res. 1999 Mar;32(3):297-301. doi: 10.1590/s0100-879x1999000300008. PMID 10347787
- [Background] Rodrigues ML, Costa RS, Souza CS, Foss NT, Roselino AM. Nephrotoxicity attributed to meglumine antimoniate (Glucantime) in the treatment of generalized cutaneous leishmaniasis. Rev Inst Med Trop Sao Paulo. 1999 Jan-Feb;41(1):33-7. doi: 10.1590/s0036-46651999000100007. PMID 10436668
- [Background] Sampaio RN, de Paula CD, Sampaio JH, Furtado Rde S, Leal PP, Rosa TT, Rodrigues ME, Veiga JP. [The evaluation of the tolerance and nephrotoxicity of pentavalent antimony administered in a dose of 40 mg Sb V/kg/day, 12/12 hr, for 30 days in the mucocutaneous form of leishmaniasis]. Rev Soc Bras Med Trop. 1997 Nov-Dec;30(6):457-63. doi: 10.1590/s0037-86821997000600003. Portuguese. PMID 9463192
- [Background] Schubach Ade O, Marzochi KB, Moreira JS, Schubach TM, Araujo ML, Vale AC, Passos SR, Marzochi MC. Retrospective study of 151 patients with cutaneous leishmaniasis treated with meglumine antimoniate. Rev Soc Bras Med Trop. 2005 May-Jun;38(3):213-7. doi: 10.1590/s0037-86822005000300001. Epub 2005 May 4. PMID 15895170
- [Background] Sharquie KE. A new intralesional therapy of cutaneous leishmaniasis with hypertonic sodium chloride solution. J Dermatol. 1995 Oct;22(10):732-7. doi: 10.1111/j.1346-8138.1995.tb03911.x. PMID 8586751
- [Background] Veiga JP, Wolff ER, Sampaio RN, Marsden PD. Renal tubular dysfunction in patients with mucocutaneous leishmaniasis treated with pentavalent antimonials. Lancet. 1983 Sep 3;2(8349):569. doi: 10.1016/s0140-6736(83)90595-0. No abstract available. PMID 6136717